CLINICAL TRIAL: NCT06100250
Title: Zenyth: Feasibility and Acceptability of an Motivational Interviewing (MI)-Based Telehealth Intervention for Bacterial Sexually Transmitted Infection (STI) Screening
Brief Title: Zenyth: Motivational Interviewing-based Telehealth Intervention for Bacterial Sexually Transmitted Infection Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Akshay Sharma, Associate Professor, University of Michigan School of Nursing, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00240181; 1R21AI168606-01A1 (NIH)
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Sexually Transmitted Diseases; Gonorrhea; Chlamydia; Syphilis; HIV
Keywords: Specimen Collection; Audio/Video Conferencing; Motivational Interviewing; Sexual and Gender Minorities; Telemedicine
MeSH Terms: conditions — Sexually Transmitted Diseases; Gonorrhea; Chlamydia Infections; Syphilis; Coitus | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth intervention (Experimental): Participants will receive an MI-based telehealth intervention for bacterial STI screening.
  Interventions: Behavioral: Motivational interviewing and specimen self-collection

INTERVENTIONS:
Behavioral: Motivational interviewing and specimen self-collection — Participants will be asked to attend a pre-test live AV conferencing session, collect and return a urine sample, a throat swab, a rectal swab, and a blood sample for bacterial STI testing, and attend a post-test live AV conferencing session.

SUMMARY:
In the United States (US), gay and bisexual men living with human immunodeficiency virus (HIV) bear a heavy burden of bacterial sexually transmitted infections (STIs) such as gonorrhea, chlamydia, and syphilis. It is important to diagnose and treat STIs in a timely manner to prevent health complications and reduce transmissions. The purpose of this study is to understand whether gay and bisexual men living with HIV are willing to collect and return specimens for bacterial STI testing when combined with live audio/video (AV) conferencing support.

DETAILED DESCRIPTION:
Participants will be recruited from across the US via social media advertising and peer referral. Seventy-five participants that complete an online survey (called the baseline survey) will be asked to attend a pre-test live AV conferencing session, collect and return a urine sample, a throat swab, a rectal swab, and a blood sample for bacterial STI testing, attend a post-test live AV conferencing session, and complete another online survey (called the satisfaction survey). Some participants (20 of 75) will also be invited to attend an online interview to share study-related experiences.

ELIGIBILITY:
Inclusion Criteria:

* Individual self-reports identifying as a man (regardless of sex assigned at birth) in the eligibility screener
* Individual self-reports residing in a US state or territory in the eligibility screener
* Individual self-reports being physically located in a US state or territory when completing study activities in the eligibility screener
* Individual self-reports being greater than or equal to (≥)18 years of age in the eligibility screener
* Individual self-reports being of legal age to provide consent for research participation in the US state or territory of residence in the eligibility screener
* Individual self-reports having been diagnosed with HIV in the eligibility screener
* Individual self-reports having any kind of condomless sex (e.g., oral, anal) with ≥2 men in the past year in the eligibility screener
* Individual self-reports being willing to provide contact information (full name, email address, mobile phone number, and mailing address) in the eligibility screener
* Individual self-reports being able to participate in live AV conferencing sessions using an internet-connected device (e.g., computer, tablet, smartphone) in the eligibility screener
* Individual self-reports being willing to receive a box that contains kits to self-collect a urine sample, a throat swab, a rectal swab, and a blood sample for bacterial STI testing in the eligibility screener
* Individual provides valid contact information (full name, email address, mobile phone number, and mailing address) in the contact information form
* Individual completes the baseline survey in order to receive the intervention

Exclusion Criteria:

* Individual self-reports not identifying as a man (regardless of sex assigned at birth) in the eligibility screener
* Individual self-reports not residing in a US state or territory in the eligibility screener
* Individual self-reports not being physically located in a US state or territory when completing study activities in the eligibility screener
* Individual self-reports not being ≥18 years of age in the eligibility screener
* Individual self-reports not being of legal age to provide consent for research participation in the US state or territory of residence in the eligibility screener
* Individual self-reports not having been diagnosed with HIV in the eligibility screener
* Individual self-reports not having any kind of condomless sex (e.g., oral, anal) with ≥2 men in the past year in the eligibility screener
* Individual self-reports not being willing to provide contact information (full name, email address, mobile phone number, and mailing address) in the eligibility screener
* Individual self-reports not being able to participate in live AV conferencing sessions using an internet-connected device (e.g., computer, tablet, smartphone) in the eligibility screener
* Individual self-reports not being willing to receive a box that contains kits to self-collect a urine sample, a throat swab, a rectal swab, and a blood sample for bacterial STI testing in the eligibility screener
* Individual does not provide valid contact information (full name, email address, mobile phone number, and mailing address) in the contact information form
* Individual does not complete the baseline survey in order to receive the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individual self-reports identifying as a man (regardless of sex assigned at birth)
Enrollment: 75 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Sharma, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Study results will be publicly reported through presentations at domestic and international conferences, and publications in peer-reviewed journals. Once analyses relating to the major aims of the proposed study have been completed and reported, the data will be deposited with the Inter-university Consortium for Political and Social Research (ICPSR) located at the University of Michigan. All confidentiality requirements will be followed as outlined on the website. ICPSR will make the data available to over 750 universities, government agencies, and other institutions, permitting other researchers to conduct secondary analyses. Data availability will be announced on the ICPSR website.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available within 6 months after analyses relating to the major aims of the proposed study have been completed and reported, and will remain available for at least 5 years.
Access Criteria: Creating an account on the ICPSR website.
URL: https://www.icpsr.umich.edu/web/pages/

REFERENCES:
- [Derived] Sharma A, Boyd S, Bonar EE. Feasibility and Acceptability of a Motivational Interviewing-Based Telehealth Intervention for Bacterial Sexually Transmitted Infection Screening: Protocol for a Sequential Explanatory Mixed Methods Study. JMIR Res Protoc. 2024 Aug 29;13:e64433. doi: 10.2196/64433. PMID 39208425

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between April 2024 and October 2024 via advertising on mobile dating apps and social networking sites.
Groups:
- Telehealth Intervention: Participants received an MI-based telehealth intervention for bacterial STI screening. Participants were asked to attend a pre-test live AV conferencing session, collect and return a urine sample, a throat swab, a rectal swab, and a blood sample for bacterial STI testing, and attend a post-test live AV conferencing session
Period: Overall Study
Arm/Group | Telehealth Intervention
Started | 75
Completed | 70
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.91 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 43
  More than one race | 5
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Schedule a Pre-test Session
Time Frame: Up to 8 weeks after participants complete the baseline survey
Population: Analysis population includes all 75 participants who were invited to schedule a pre-test session after completing the baseline survey
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 75
Participants | 74

2. Primary Outcome: Number of Participants That Join the Pre-test Session Within 30 Minutes of the Start Time
Time Frame: Up to 8 weeks after participants complete the baseline survey
Population: Analysis population only includes 74 participants who actually scheduled a pre-test session after being invited
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 74
Participants | 69

3. Primary Outcome: Number of Participants That Return Each Type of Specimen Within 6 Weeks of Box Delivery
Time Frame: Up to 16 weeks after participants complete the baseline survey
Population: Analysis population only includes 69 participants who were shipped a specimen self-collection box after completing the pre-test session
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 69
Participants
  Urine sample | 57
  Throat swab | 57
  Rectal swab | 57
  Blood sample | 54

4. Primary Outcome: Number of Participants That Provide Specimens of Adequate Quality for Lab Testing
Time Frame: Up to 16 weeks after participants complete the baseline survey
Population: Analysis population only includes 57 participants who returned at least one type of specimen after receiving the specimen self-collection box
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 57
Participants
  Urine sample | 57
  Throat swab | 56
  Rectal swab | 55
  Blood sample: number analyzed (Participants) | 54
  Blood sample | 47

5. Primary Outcome: Number of Participants That Schedule a Post-test Session
Time Frame: Up to 24 weeks after participants complete the baseline survey
Population: Analysis population only includes 57 participants who were invited to schedule a post-test session after returning at least one type of specimen
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 57
Participants | 57

6. Primary Outcome: Number of Participants That Join the Post-test Session Within 30 Minutes of the Start Time
Time Frame: Up to 24 weeks after participants complete the baseline survey
Population: Analysis population only includes 57 participants who actually scheduled a post-test session after being invited
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 57
Participants | 55

7. Primary Outcome: Overall Intervention Satisfaction
Description: Participants' satisfaction with the pre-test session, urine sample collection, throat swab collection, rectal swab collection, blood sample collection, and the post-test session will be assessed using six 5-point Likert items included in the satisfaction survey. Response values will be summed to obtain a total score ranging from 6-30, with higher scores indicating greater overall intervention satisfaction.
Time Frame: Up to 32 weeks after participants complete the baseline survey
Population: Analysis population only includes 47 participants who answered the questions on satisfaction with the pre-test session, urine sample collection, throat swab collection, rectal swab collection, blood sample collection, and the post-test session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 47
score on a scale | 28.09 (2.42)

8. Primary Outcome: Interventionist Perceptions
Description: Participants' perceptions of the interventionist conducting the pre-test and the post-test sessions will be assessed using two 12-item Counselor Rating Form Short scales included in the satisfaction survey. Response values will be summed to obtain a total score ranging from 24-168, with higher scores indicating more positive interventionist perceptions.
Time Frame: Up to 32 weeks after participants complete the baseline survey
Population: Analysis population only includes 51 participants who answered the questions on perceptions of the interventionist conducting the pre-test and the post-test sessions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 51
score on a scale | 163.92 (20.39)

9. Primary Outcome: Usability of the Pre-test and the Post-test Sessions
Description: Participants' usability of the pre-test and the post-test sessions will be assessed using two 4-item subscales from the Telehealth Usability Questionnaire on the quality of interactions with the interventionist during each session included in the satisfaction survey. Response values will be summed to obtain a total score ranging from 8-56, with higher scores indicating greater usability of the pre-test and the post-test sessions.
Time Frame: Up to 32 weeks after participants complete the baseline survey
Population: Analysis population only includes 52 participants who answered the questions on usability of the pre-test and the post-test sessions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 52
score on a scale | 53.56 (7.14)

10. Primary Outcome: Willingness to Repeat the Intervention
Description: Participants' willingness to repeat the pre-test session, urine sample collection, throat swab collection, rectal swab collection, blood sample collection, and the post-test session will be assessed using six 5-point Likert items included in the satisfaction survey. Response values will be summed to obtain a total score ranging from 6-30, with higher scores indicating greater willingness to repeat the intervention.
Time Frame: Up to 32 weeks after participants complete the baseline survey
Population: Analysis population only includes 48 participants who answered the questions on willingness to repeat the pre-test session, urine sample collection, throat swab collection, rectal swab collection, blood sample collection, and the post-test session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 48
score on a scale | 28.60 (2.32)

11. Primary Outcome: Likelihood of Recommending the Intervention to Friends or Sex Partners
Description: Participants' likelihood of recommending the pre-test session, urine sample collection, throat swab collection, rectal swab collection, blood sample collection, and the post-test session to friends or sex partners will be assessed using six 5-point Likert items included in the satisfaction survey. Response values will be summed to obtain a total score ranging from 6-30, with higher scores indicating greater likelihood of recommending the intervention to friends or sex partners.
Time Frame: Up to 32 weeks after participants complete the baseline survey
Population: Analysis population only includes 46 participants who answered the questions on likelihood of recommending the pre-test session, urine sample collection, throat swab collection, rectal swab collection, blood sample collection, and the post-test session to friends or sex partners
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 46
score on a scale | 28.33 (2.30)

12. Secondary Outcome: Change in STI-related Knowledge
Description: Potential changes in participants' knowledge of gonorrhea, chlamydia, and syphilis will be assessed by comparing responses to the same set of 22 items included in the baseline survey and the satisfaction survey. Response values will be summed to obtain separate total scores ranging from 0-22, with higher scores indicating greater STI-related knowledge. A positive value for the difference in scores (post-test minus pre-test) represents an increase, and a negative value for the difference in scores (post-test minus pre-test) represents a decrease.
Time Frame: Pre-intervention score (from the baseline survey); Post-intervention score (from the satisfaction survey completed up to 32 weeks after participants complete the baseline survey)
Population: Analysis population only includes 67 participants who answered the questions assessing knowledge of gonorrhea, chlamydia, and syphilis in the baseline survey and the satisfaction survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 67
score on a scale
  Pre-intervention score (from the baseline survey) | 16.34 (3.48)
  Post-intervention score (from the satisfaction survey) | 17.16 (3.41)
  Difference | 0.82 (2.66)
Statistical Analysis 1: Comparison: Telehealth Intervention; Null hypothesis = Mean difference between the paired STI-related knowledge scores (pre-intervention and post-intervention) is 0; Test type: Other — Paired sample t-test, 2 sided; p = 0.01, Paired sample t-test, 2 sided — A priori threshold for statistical significance = 0.05; Degrees of freedom = 66; Mean Difference (Net) = 0.82 — Estimation parameter represents the average of the differences between the paired observations (post-intervention score minus pre-intervention score)

13. Secondary Outcome: Likelihood of Testing for Bacterial STIs at Least Annually
Description: Participants' likelihood of testing for bacterial STIs at least annually will be assessed using a single 5-point Likert item included in the satisfaction survey. Response values will range from 1-5, with higher values indicating greater likelihood of testing for bacterial STIs at least annually.
Time Frame: Up to 32 weeks after participants complete the baseline survey
Population: Analysis population only includes 70 participants who answered the question on likelihood of testing for bacterial STIs at least annually
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 70
score on a scale | 4.91 (0.37)

14. Secondary Outcome: Change in Self-efficacy for Specimen Self-collection
Description: Potential changes in participants' self-efficacy for urine sample collection, throat swab collection, rectal swab collection, and blood sample collection will be assessed by comparing responses to similar sets of four 5-point Likert items included in the baseline survey and the satisfaction survey. Response values will be summed to obtain separate total scores ranging from 4-20, with higher scores indicating greater self-efficacy for specimen self-collection. A positive value for the difference in scores (post-test minus pre-test) represents an increase, and a negative value for the difference in scores (post-test minus pre-test) represents a decrease.
Time Frame: as for outcome 12
Population: Analysis population only includes 48 participants who answered the questions assessing self-efficacy for urine sample collection, throat swab collection, rectal swab collection, and blood sample collection in the baseline survey and the satisfaction survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 48
score on a scale
  Pre-intervention score (from the baseline survey) | 18.83 (1.64)
  Post-intervention score (from the satisfaction survey) | 17.54 (2.69)
  Difference | -1.29 (2.17)
Statistical Analysis 1: Comparison: Telehealth Intervention; Null hypothesis = Mean difference between the paired self-efficacy for specimen self-collection scores (pre-intervention and post-intervention) is 0; Test type: Other — Paired sample t-test, 2 sided; p < 0.01, Paired sample t-test, 2 sided — A priori threshold for statistical significance = 0.05; Degrees of freedom = 47; Mean Difference (Net) = -1.29 — [estimate comment as in outcome 12, analysis 1]

15. Secondary Outcome: Number of Participants That Test Negative or Positive for Gonorrhea, Chlamydia, and Syphilis
Time Frame: Up to 16 weeks after participants complete the baseline survey
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 57
Participants
  Gonorrhea PCR: Negative | 43
  Gonorrhea PCR: Positive | 11
  Gonorrhea PCR: Unable to Analyze Specimen | 3
  Chlamydia PCR: Negative | 50
  Chlamydia PCR: Positive | 4
  Chlamydia PCR: Unable to Analyze Specimen | 3
  Syphilis RPR: number analyzed (Participants) | 54
  Syphilis RPR: Negative | 29
  Syphilis RPR: Positive | 18
  Syphilis RPR: Unable to Analyze Specimen | 7

16. Secondary Outcome: Number of Participants That Initiate Treatment Within 1 Week of Receiving a Positive Test Result
Time Frame: Up to 28 weeks after participants complete the baseline survey
Population: Analysis population only includes 24 participants who tested positive for gonorrhea, chlamydia, or syphilis
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Intervention
Number analyzed (Participants) | 24
Participants | 5

ADVERSE EVENTS:
Time Frame: Up to 32 weeks after participants complete the baseline survey
Arm/Group | Telehealth Intervention
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT06100250/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT06100250/ICF_002.pdf